CLINICAL TRIAL: NCT01532271
Title: Comparison of Brain Network Activation Analysis (BNA™) Using Evoked Response Potentials, Clinical Symptoms and Neuro-cognitive Performance and Symptoms in Concussed Children, Young Adults and Matched Controls
Brief Title: Comparison of Brain Network Activation (BNA™) Analysis, Clinical Symptoms and Neuro-cognitive Performance in Concussed Children and Young Adults
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-01
Record Dates: First submitted 2012-02-07; First posted 2012-02-14 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury
Keywords: mild Traumatic Brain Injury; mTBI; Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concussed: Patients with recent concussion
- Matched controls: Athletes with no recent concussion

SUMMARY:
The use of Event Related Potentials (ERP) and neurocognitive performance in patients following concussion has been examined previously in small cohorts and relatively long after concussion occurred. However, little is known about the immediate changes in brain activity in specific brain regions and connectivity across them associated with performance on specific neurocognitive tests following a concussion, and the subsequent changes over time. The proposed study will provide initial evidence for the feasibility of an ERP based biomarker for concussion reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with concussion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-27 years
* Arm 1 only (Concussed): Over 2 days and below 10 days post-concussion (sports-related)
* Currently symptomatic
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self)

Exclusion Criteria:

* TBI (i.e., Glasgow Coma Scale <13) or brain surgery
* Any psychiatric disorder
* Substance abuse
* Special education
* Any Neurological disorder
* Any medication affecting CNS
* Significant sensory deficits such as deafness or blindness
* Clinically significant abnormal laboratory values or ECG
* A history of more than 3 concussions in the past
* A concussion within the last year
* Residual symptoms or deficits related to a previous concussion

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Experimental subjects will include males and females with a recent sports-related concussion (less than 10 days post-concussion) recruited from approximately 50 high schools and colleges with UPMC-affiliated certified athletic trainers (ATC) on staff and from patients at the UPMC Sports Medicine Concussion Program.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change of Brain Network Activation(BNA™)Scores Over Post Concussion Recovery Period | days 2-10, 7-19, 12-28, 17-37 following concussion

SECONDARY OUTCOMES:
Correlation Of The Change In BNA™ Scores To Neurocognitive Tests Scores and Clinical Diagnostic | days 2-10, 7-19, 12-28, 17-37 following concussion

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P. Kontos, Ph.D., Principal Investigator — UPMC Sports Medicine Concussion Program; Michael W. Collins, Ph.D., Principal Investigator — UPMC Sports Medicine Concussion Program
Locations (1):
- UPMC Sports Medicine Concussion Program, Pittsburgh, Pennsylvania, United States